CLINICAL TRIAL: NCT03309241
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study To Assess The Safety, Tolerability, And Pharmacokinetics Of Single Escalating Oral Doses Of Pf-06882961 In Healthy Adult Subjects
Brief Title: First In Human, Single Escalating Oral Dose Study Of PF-06882961 In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: C3421001
Record Dates: First submitted 2017-10-10; First posted 2017-10-13 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — danuglipron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind (sponsor open)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Single Ascending Dose in crossover design with placebo substitution. Administration under fed or fasted conditions as tablet or solution formulation. At least 7 days washout between doses in an individual subject.
  Interventions: Drug: PF-06882961; Other: Placebo
- Cohort 2 (Experimental): Single Ascending Dose in crossover design with placebo substitution. Administration under fed or fasted conditions as tablet or solution formulation. At least 7 days washout between doses in an individual subject.
  Interventions: Drug: PF-06882961; Other: Placebo
- Cohort 3 (optional) (Experimental): Single Ascending Dose administration under fed or fasted conditions as tablet or solution formulation. At least 7 days washout between doses in an individual subject.
  Interventions: Drug: PF-06882961; Other: Placebo

INTERVENTIONS:
Drug: PF-06882961 — Single Ascending Doses of PF-06882961 from 3mg to TBD mg.
Other: Placebo — Placebo Single Dose

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of single oral doses of PF-06882961 in healthy adult subjects. This is the first clinical study of PF-06882961.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of nonchildbearing potential and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive
* Body mass index (BMI) within 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb)
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal (including pancreatitis), cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of IP (whichever is longer).
* Fertile male subjects who are unwilling or unable to use a highly effective method of contraception for the duration of the study and for at least 28 days after the last dose.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Seriousness and Relationship to Treatment | First dose of study drug up to 28 days after last dose of study drug
  Assessment by adverse event monitoring, 12 lead ECGs, cardiac telemetry, vital signs and clinical safety laboratory measurements.

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | Pre-dose and at 0.3, 0.75, 1.25,2,3,4,6,8,10,12,24,36,48 hours following single dose administration
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Maximum Observed Plasma Concentration (Cmax) | Pre-dose and at 0.3, 0.75, 1.25,2,3,4,6,8,10,12,24,36,48 hours following single dose administration
  Maximum Observed Plasma Concentration (Cmax)
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Pre-dose and at 0.3, 0.75, 1.25,2,3,4,6,8,10,12,24,36,48 hours following single dose administration
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Plasma Decay Half-Life (t1/2) | Pre-dose and at 0.3, 0.75, 1.25,2,3,4,6,8,10,12,24,36,48 hours following single dose administration
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C3421001&StudyName=A+Phase+1%2C+Randomized%2C+Double+Blind%2C+Placebo+Controlled+Study+To+Assess+The+Safety%2C+Tolerability%2C+And+Pharmacokinetics+Of+Single+Escalating+Oral+Doses+Of+Pf+06882961+In+Healthy+Adult+Subjects
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C3421001&StudyName=A+Phase+1%2C+Randomized%2C+Double-blind%2C+Placebo-controlled+Study+To+Assess+The+Safety%2C+Tolerability%2C+And+Pharmacokinetics+Of+Single+Escalating+Oral+Doses+Of+Pf-06882961+In+Healthy+Adult+Subjects